CLINICAL TRIAL: NCT01726023
Title: A Phase III, Randomized, Multicenter, Double Blind, Double-Dummy, Parallel-Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-Abdominal Infections In Hospitalized Adults
Brief Title: Compare Ceftazidime-Avibactam + Metronidazole vs Meropenem for Hospitalized Adults With Complicated Intra-Abd Infections
Acronym: RECLAIM3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4280C00018; 2011-003893-97
Record Dates: First submitted 2012-11-05; First posted 2012-11-14 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Complicated Intra-abdominal Infection
Keywords: Ceftazidime-avibactam,; Metronidazole,; Meropenem,; Anti-Bacterial Agents,; Anti-Infective Agents,; Therapeutic Uses,; Pharmacologic Actions,; Physiological Effects of Drugs
MeSH Terms: interventions — avibactam, ceftazidime drug combination; Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ceftazidime-Avibactam plus metronidazole (Experimental)
  Interventions: Drug: Ceftazidime-avibactam; Drug: metronidazole
- Meropenem (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Ceftazidime-Avibactam powder for concentrate for solution for infusion 2000 mg/500 mg
  Arms: Ceftazidime-Avibactam plus metronidazole
Drug: metronidazole — Metronidazole 500mg/100ml solution for infusion
  Arms: Ceftazidime-Avibactam plus metronidazole
Drug: Meropenem — Meropenem powder for solution for infusion 1000mg
  Arms: Meropenem

SUMMARY:
The purpose of this study is to evaluate the effects of Ceftazidime Avibactam plus Metronidazole compared to Meropenem for treating hospitalized patients with complicated intra-abdominal infections.

DETAILED DESCRIPTION:
A Phase III, Randomized, Multicenter, Double Blind, Double-Dummy, Parallel-Group, Comparative Study to Determine the Efficacy, Safety, and Tolerability of Ceftazidime Avibactam Plus Metronidazole Versus Meropenem in the Treatment of Complicated Intra-Abdominal Infections In Hospitalized Adults

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 to 90 years of age, inclusive,
* Female patients can participate if they are surgically sterilized or postmenopausal for at least 1 year or her sexual partner has had a vasectomy
* Female of childbearing potential has had normal menstrual periods for 3 months and negative serum pregnancy test and agree to practice highly effective methods of birth control during treatment and for at least 7 days after last dose
* Intraoperative/postoperative enrollment with visual confirmation (presence of pus within the abdominal cavity) of an intra-abdominal infection associated with peritonitis
* Confirmation of infection by surgical intervention within 24 hours of entry: evidence of systemic inflammatory indicators; physical findings consistent with intra-abdominal infection; supportive radiologic imaging findings of intra-abdominal infections

Exclusion Criteria:

* Patient is diagnosed with traumatic bowel perforation undergoing surgery within 12 hours; perforation of gastroduodenal ulcers undergoing surgery within 24 hours. Other intra-abdominal processes in which primary etiology is not likely to be infectious
* Patient has abdominal wall abscess or bowel obstruction without perforation or ischemic bowel without perforation
* Patients whose surgery will include staged abdominal repair, or "open abdomen" technique, or marsupialization
* Patient has suspected intra-abdominal infections due to fungus, parasites, virus or tuberculosis
* Patient is considered unlikely to survive the 6- to 8-week study period or has a rapidly progressive or terminal illness, including septic shock that is associated with a high risk of mortality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newell, MBBS, MRCP, Study Director — AstraZeneca
Locations (30):
- China (19):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Haikou
  - Research Site, Hebei
  - Research Site, Jiangyin
  - Research Site, Liaocheng
  - Research Site, Nanchang
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuxi
  - Research Site, Xi'an
- South Korea (9):
  - Research Site, Ansan-si
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Wŏnju
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Torres A, Wible M, Tawadrous M, Irani P, Stone GG, Quintana A, Debabov D, Burroughs M, Bradford PA, Kollef M. Efficacy and safety of ceftazidime/avibactam in patients with infections caused by beta-lactamase-producing Gram-negative pathogens: a pooled analysis from the Phase 3 clinical trial programme. J Antimicrob Chemother. 2023 Nov 6;78(11):2672-2682. doi: 10.1093/jac/dkad280. PMID 37700689
- [Derived] Cheng K, Newell P, Chow JW, Broadhurst H, Wilson D, Yates K, Wardman A. Safety Profile of Ceftazidime-Avibactam: Pooled Data from the Adult Phase II and Phase III Clinical Trial Programme. Drug Saf. 2020 Aug;43(8):751-766. doi: 10.1007/s40264-020-00934-3. PMID 32602065
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279
- [Derived] Stone GG, Newell P, Gasink LB, Broadhurst H, Wardman A, Yates K, Chen Z, Song J, Chow JW. Clinical activity of ceftazidime/avibactam against MDR Enterobacteriaceae and Pseudomonas aeruginosa: pooled data from the ceftazidime/avibactam Phase III clinical trial programme. J Antimicrob Chemother. 2018 Sep 1;73(9):2519-2523. doi: 10.1093/jac/dky204. PMID 29912399
- [Derived] Qin X, Tran BG, Kim MJ, Wang L, Nguyen DA, Chen Q, Song J, Laud PJ, Stone GG, Chow JW. A randomised, double-blind, phase 3 study comparing the efficacy and safety of ceftazidime/avibactam plus metronidazole versus meropenem for complicated intra-abdominal infections in hospitalised adults in Asia. Int J Antimicrob Agents. 2017 May;49(5):579-588. doi: 10.1016/j.ijantimicag.2017.01.010. Epub 2017 Mar 29. PMID 28363526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 486 patients were enrolled from 43 centers in 3 countries in this study. The first patient was enrolled on 14 January 2013 and the last patient last visit was on 14 March 2015.
Pre-assignment Details: Of 486 enrolled patients, 42 did not meet the eligibility criteria. A further two patients were not randomized due to withdrawn consent, and one patient was not randomized due to unavailability of study drug.
Groups:
- Ceftazidime-Avibactam Plus Metronidazole: Ceftazidime-Avibactam powder for concentrate for solution for infusion 2000 mg/500 mg Plus Metronidazole 500mg/100ml solution for infusion
Period: Overall Study
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Started | 219 | 222
Completed | 190 | 196
Not Completed | 29 | 26
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 5 | 10
Not completed — Other Eligibility criteria | 7 | 7
Not completed — Withdrawal by Subject | 16 | 8

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is MITT ; Randomized patients who received any amount of study therapy, excluding patients who received both study therapies. 9 patients were randomized but not treated, and one patient received doses of both treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem | Total
Number analyzed (Participants) | 214 | 217 | 431
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (16.83) | 48.5 (17.43) | 48.5 (17.11)
Age, Customized [Number; unit: Participants]
  18-45 Years | 89 | 96 | 185
  46-64 Years | 85 | 72 | 157
  65-74 Years | 28 | 30 | 58
  75-90 Years | 12 | 19 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 64 | 137
  Male | 141 | 153 | 294
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 214 | 217 | 431

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Clinical Cure at the Test of Cure (TOC) Visit in the Clinically Evaluable (CE) Analysis Set.
Description: The proportion of patients meeting the cure criteria: complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy, drainage, or surgical intervention was necessary.
Time Frame: At the test of cure visit (Day 28 to35)
Population: The clinically evaluable (CE) analysis set included all patients who met the disease definition of cIAI and met the stringent criteria for clinical evaluation described in the protocol regarding dosing, concomitant medication, evaluation, etc.
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 177 | 184
Number of patients
  Clinical cure | 166 | 173
  Clinical failure | 11 | 11
Statistical Analysis 1: Comparison: Ceftazidime-Avibactam Plus Metronidazole vs Meropenem; The Primary objective of this study was to assess the non inferiority (based on a 12.5% margin) of CAZ AVI plus metronidazole compared to meropenem alone with respect to clinical cure at the TOC visit in patients who were CE; Test type: Non-Inferiority or Equivalence — The non-inferiority would be concluded if the lower limit of the 95% confidence interval (CI; corresponding to a 97.5% 1 sided lower bound) was greater than -12.5% for the primary outcome variable; p < 0.001, % Risk Difference (RD) — P-value for 1-sided test at test of cure (TOC) with a -12.5% non-inferiority margin, i.e. H0: diff ≤ -12.5%; RD is CAZ AVI clinical cure rate minus Meropenem clinical cure rate. The CI was calculated by Miettinen and Nurminen method without adjustment; Risk Difference (RD) = -0.20, 95% CI 2-sided [-5.53 to 4.97] — units for RD are %

2. Secondary Outcome: The Proportion of Patients With Clinical Cure at the End of Treatment (EOT) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: Microbiologically evaluable (ME) analysis set defined as all patients included in the clinically evaluable (CE) set with at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture that was susceptible to both treatment groups.
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 106 | 118
Number of patients
  Clinical cure | 103 | 113
  Clinical failure | 3 | 5

3. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Test of Cure (TOC) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 99 | 113
Number of patients
  Clinical cure | 92 | 107
  Clinical failure | 7 | 6

4. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Late Follow up (LFU) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 96 | 106
Number of patients
  Clinical cure | 89 | 100
  Clinical failure | 7 | 6

5. Secondary Outcome: The Proportion of Patients With Clinical Cure at the End of Treatment (EOT) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: Extended microbiologically evaluable (ME) analysis set defined as all patients included in the clinically evaluable (CE) set with at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture regardless of susceptibility.
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 107 | 125
Number of patients
  Clinical cure | 104 | 120
  Clinical failure | 3 | 5

6. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Test of Cure (TOC) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 5
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 100 | 119
Number of patients
  Clinical cure | 93 | 113
  Clinical failure | 7 | 6

7. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Late Follow up (LFU) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 1
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 5
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 97 | 112
Number of patients
  Clinical cure | 90 | 106
  Clinical failure | 7 | 6

8. Secondary Outcome: The Proportion of Patients With Clinical Cure at the End of Treatment (EOT) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 1
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: The microbiological modified intent-to-treat mMITT analysis set included all randomized patients who met the disease definition of cIAI and had at least 1 etiologic pathogen identified at study entry (regardless of isolate susceptibilities). Patients with a bacterial species typically not expected to respond to both study drugs were excluded.
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Clinical cure | 126 | 140
  Clinical failure | 6 | 7
  Indeterminate | 11 | 5

9. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Test of Cure (TOC) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 1
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 8
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Clinical cure | 119 | 135
  Clinical failure | 10 | 9
  Indeterminate | 14 | 8

10. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Late Follow up (LFU) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 1
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 8
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Clinical cure | 116 | 132
  Clinical failure | 10 | 9
  Indeterminate | 17 | 11

11. Secondary Outcome: The Proportion of Patients With Clinical Cure at the End of Treatment (EOT) Visit in the Clinically Evaluable (CE) Analysis Set.
Description: as for outcome 1
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 190 | 196
Number of patients
  Clinical cure | 183 | 187
  Clinical failure | 7 | 9

12. Secondary Outcome: The Proportion of Patients With Clinical Cure at the Late Follow up (LFU) Visit in the Clinically Evaluable (CE) Analysis Set.
Description: as for outcome 1
Time Frame: At late follow up (LFU) visits (Day 42 to 49)
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 168 | 179
Number of patients
  Clinical cure | 157 | 168
  Clinical failure | 11 | 11

13. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the End of Treatment (EOT) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: Per-patient "favorable" response indicates that all of the patient's baseline pathogens are "eradicated" or "presumed eradicated".
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 106 | 118
Number of patients
  Favorable | 103 | 113
  Unfavorable | 3 | 5

14. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Test of Cure (TOC) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 13
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 99 | 113
Number of patients
  Favorable | 92 | 107
  Unfavorable | 7 | 6

15. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Late Follow up (LFU) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 13
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 96 | 106
Number of patients
  Favorable | 89 | 100
  Unfavorable | 7 | 6

16. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the End of Treatment (EOT) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 13
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: as for outcome 5
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 107 | 125
Number of patients
  Favorable | 104 | 120
  Unfavorable | 3 | 5

17. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Test of Cure (TOC) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 13
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 5
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 100 | 119
Number of patients
  Favorable | 93 | 113
  Unfavorable | 7 | 6

18. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Late Follow up (LFU) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 13
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 5
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 97 | 112
Number of patients
  Favorable | 90 | 106
  Unfavorable | 7 | 6

19. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the End of Treatment (EOT) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 13
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all randomized patients who met the disease definition of cIAI and had at least 1 etiologic pathogen identified at study entry (regardless of isolate susceptibilities). Patients with a bacterial species typically not expected to respond to both study drugs were excluded.
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Favorable | 126 | 140
  Unfavorable | 6 | 7
  Indeterminate | 11 | 5

20. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Test of Cure (TOC) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 13
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 19
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Favorable | 119 | 135
  Unfavorable | 10 | 9
  Indeterminate | 14 | 8

21. Secondary Outcome: The Proportion of Patients With a Favorable Per-patient Microbiological Response at the Late Follow up (LFU) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 13
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 19
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Number of patients
  Favorable | 116 | 132
  Unfavorable | 10 | 9
  Indeterminate | 17 | 11

22. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the End of Treatment (EOT) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: The proportion of patients with a favorable per-pathogen microbiological response: favourable microbiological response includes: Eradication Absence of causative pathogen from specimens at the site of infection. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure.
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: The mMITT analysis set included all randomized patients who met the disease definition of cIAI and had at least 1 etiologic pathogen identified at study entry (regardless of isolate susceptibilities). Patients with a bacterial species typically not expected to respond to both study drugs were excluded.
Measure: Number; unit: Participants with favorable responses
Groups:
- Ceftazidime-Avibactam Plus Metronidazole: Ceftazidime-Avibactam powder for concentrate for solution for infusion 2000 mg/500 mg Plus Metronidazole 500mg/100ml solution for infusion (summary only shows pathogens where N>/=10)
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Participants with favorable responses
  Escherichia coli (n=84, 89) | 77 | 86
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=28,35) | 22 | 32
  Pseudomonas aeruginosa (n=17, 20) | 15 | 17
  Streptococcus anginosus grou (n=8, 7) | 7 | 6
  Streptococcus mitis group (n=6, 5) | 6 | 5
  Enterococcus faecalis (n=6, 6) | 5 | 5
  Enterococcus faecium (n=4, 7) | 4 | 5

23. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response in the Microbiological Response at the Test of Cure (TOC) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 22
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 22
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Participants with favorable responses
  Escherichia coli (n=84, 89) | 70 | 84
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=28,35) | 23 | 31
  Pseudomonas aeruginosa (n=17, 20) | 14 | 17
  Streptococcus anginosus group (n=8, 7) | 7 | 5
  Streptococcus mitis group (n=6, 5) | 6 | 5
  Enterococcus faecalis (n=6, 6) | 6 | 4
  Enterococcus faecium (n=4, 7) | 4 | 5

24. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response in the Microbiological Response at the Late Follow up (LFU) Visit in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: as for outcome 22
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 22
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 143 | 152
Participants with favorable responses
  Escherichia coli (n=84, 89) | 70 | 82
  Klebsiella pneumoniae (n=28, 35) | 22 | 31
  Pseudomonas aeruginosa (n=17, 20) | 14 | 17
  Klebsiella oxytoca (n=5, 5) | 4 | 5
  Enterococcus faecalis (n=6, 6) | 4 | 4
  Enterococcus faecium (n=4, 7) | 3 | 5
  Streptococcus anginosus group (n=8, 7) | 7 | 5
  Streptococcus mitis group (n=6, 5) | 6 | 5

25. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the End of Treatment (EOT) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: as for outcome 2
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 99 | 113
Participants with favorable responses
  Escherichia coli (n=69, 77) | 68 | 75
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=22, 29) | 21 | 28
  Pseudomonas aeruginosa (n=14, 16) | 14 | 14

26. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the Test of Cure (TOC) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 2
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 99 | 113
Participants with favorable responses
  Escherichia coli (n=69, 77) | 64 | 74
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=22, 29) | 21 | 28
  Pseudomonas aeruginosa (n=14, 16) | 13 | 14

27. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the Late Follow up (LFU) Visit in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 2
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 99 | 113
Participants with favorable responses
  Escherichia coli (n=69, 77) | 63 | 72
  Klebsiella oxytoca (n=5, 5) | 4 | 5
  Klebsiella pneumoniae (n=22, 29) | 21 | 27
  Pseudomonas aeruginosa (n=14, 16) | 13 | 14

28. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the End of Treatment (EOT) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the end of treatment (EOT) (within 24 hours after last IV dose)
Population: Extended microbiologically evaluable(ME) analysis set defined as all patients included in the clinically evaluable (CE) set with at least 1 Gram-negative aerobic pathogen in the initial/prestudy culture regardless of susceptibility.
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 100 | 119
Participants with favorable responses
  Escherichia coli (n=70, 80) | 69 | 78
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=22, 30) | 21 | 29
  Pseudomonas aeruginosa (n=14, 18) | 14 | 16

29. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the Test of Cure (TOC) Visit in the Extended Microbiologically Evaluable(ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 28
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 100 | 119
Participants with favorable responses
  Escherichia coli (n=70, 80) | 65 | 77
  Klebsiella oxytoca (n=5, 5) | 5 | 5
  Klebsiella pneumoniae (n=22, 30) | 21 | 29
  Pseudomonas aeruginosa (n=14, 18) | 13 | 16

30. Secondary Outcome: The Proportion of Favorable Per-pathogen Microbiological Response at the Late Follow up (LFU) Visit in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 22
Time Frame: At the late follow up (LFU) (Day 42 to 49)
Population: as for outcome 28
Measure: Number; unit: Participants with favorable responses
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 100 | 119
Participants with favorable responses
  Escherichia coli (n=70, 80) | 64 | 75
  Klebsiella oxytoca (n=5, 5) | 4 | 5
  Klebsiella pneumoniae (n=22, 30) | 21 | 28
  Pseudomonas aeruginosa (n=14, 18) | 13 | 16

31. Secondary Outcome: The Proportion of Patients With a Favorable Per Patient Microbiological Response at the Test of Cure (TOC) Visit for Patients Infected With Ceftazidime Resistant Pathogens in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set.
Description: The microbiological responses as per the protocoled criteria: responses other than "indeterminate" were classified as "favorable" or "unfavorable." Favorable microbiological response assessments included "eradication" and "presumed eradication." Unfavorable microbiological response assessments included "persistence," "persistence with increasing minimum inhibitory concentration (MIC)," and "presumed persistence." Indeterminate microbiologic response assessments included cases where the clinical response was changed to indeterminate due to an SRP assessment of inadequate source control (ie, circumstances that preclude classification as eradication, presumed eradication, persistence, persistence with increasing MIC, and presumed persistence).
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 19
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 29 | 29
Number of patients
  Favorable | 24 | 27
  Unfavorable | 1 | 1
  Indeterminate | 4 | 1

32. Secondary Outcome: The Proportion of Patients With a Favorable Per Patient Microbiological Response at the Test of Cure (TOC) Visit for Patients Infected With Ceftazidime Resistant Pathogens in the Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 31
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 2
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 23 | 24
Number of patients
  Favorable | 22 | 23
  Unfavorable | 1 | 1

33. Secondary Outcome: The Proportion of Patients With a Favorable Per Patient Microbiological Response at the Test of Cure (TOC) Visit for Patients Infected With Ceftazidime Resistant Pathogens in the Extended Microbiologically Evaluable (ME) Analysis Set.
Description: as for outcome 31
Time Frame: At the test of cure (TOC) (Day 28 to 35)
Population: as for outcome 28
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 23 | 26
Number of patients
  Favorable | 22 | 25
  Unfavorable | 1 | 1

34. Secondary Outcome: The Time to First Defervescence in the Clinically Evaluable (CE) Analysis Set for Patients Who Have Fever at Study Entry.
Description: Time to first defervescence was calculated for patients with a fever (>38ºC) at baseline. Defervescence (≤37.8ºC) was defined as the absence of fever based on the highest temperature recorded on each study day. Time to first defervescence while on IV study therapy in the CE analysis set at TOC for patients who had fever at study entry is defined as time (in days) from the first dose of IV study therapy to first absence of fever.
Time Frame: while on study therapy (from Day 1 to Day 14)
Population: Clinically evaluable (CE) with fever, defined as >38ºC at study entry. No participants were censored at the time of last observation.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 17 | 26
Days | 1 [1 to 5] | 1.5 [1 to 4]
Statistical Analysis 1: Comparison: Ceftazidime-Avibactam Plus Metronidazole vs Meropenem; Test type: Superiority or Other; p = 0.773, Log Rank; Difference in median time (days) = 0.5

35. Secondary Outcome: The Time to First Defervescence in the Microbiological Modified Intent-to-treat (mMITT) Analysis Set for Patients Who Have Fever at Study Entry.
Description: as for outcome 34
Time Frame: while on study therapy (from Day 1 to Day 14)
Population: microbiological modified intent-to-treat (mMITT) with fever, defined as >38ºC at study entry. No participants were censored at the time of last observation.
Measure: Median (Full Range); unit: Days
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 16 | 26
Days | 1 [1 to 5] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Ceftazidime-Avibactam Plus Metronidazole vs Meropenem; Test type: Superiority or Other; p = 0.598, Log Rank; Difference in median time (days) = 1

36. Secondary Outcome: Safety and Tolerability by Incidence and Severity of Adverse Events and Serious Adverse Events and Mortality.
Description: Adverse event data were collected from the screening/consent visit until the late follow-up visit (i.e. Day -1/0 to Day 42).
Time Frame: study duration (from screening to Day 49 LFU visit)
Population: Safety analysis set: all patients who received at least 1 dose of IP
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 215 | 217
Number of patients
  Any AE | 82 | 83
  Any SAE | 9 | 11
  Any AE leading to discontinuation of IP | 7 | 3
  Any AE of severe intensity | 5 | 5
  Total number of deaths | 2 | 1
  Deaths due to disease progression | 2 | 0
  Any AE with outcome=death | 0 | 1

37. Secondary Outcome: Safety and Tolerability by Incidence: Extent of Exposure.
Description: Duration of exposure is calculated as the difference between the last study therapy date and the first study therapy date converted to days plus 1 day. Actual calculated duration could be shorter or longer than a full day.
Time Frame: study duration (from screening to Day 49 LFU visit)
Population: Safety analysis set: all patients who received at least 1 dose of IP
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 215 | 217
Number of patients
  1 - 2 days | 10 | 5
  3 - 4 days | 6 | 5
  5 -10 days | 175 | 181
  11 - 14 days | 24 | 26
  >14 days | 0 | 0

38. Secondary Outcome: Safety and Tolerability: Clinical Laboratory Evaluation Hematology.
Description: Potentially clinically significant (PCS) post Baseline hematology values up to LFU (Safety analysis set)
Time Frame: study duration (from screening to Day 49 LFU visit)
Population: Safety analysis set: all patients who received at least 1 dose of IP
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 215 | 217
Number of patients
  Platelet count: PCS (Low) | 1 | 1
  Platelet count: PCS (High) | 5 | 4
  Red blood cell count: PCS (Low) | 7 | 13
  Red blood cell count: PCS (High) | 0 | 0
  White blood cell: PCS (Low) | 1 | 1
  White blood cell: PCS (High) | 4 | 5
  Hemoglobin: PCS (Low) | 7 | 14
  Hemoglobin: PCS (High) | 0 | 0
  Lymphocytes: PCS (Low) | 1 | 1
  Lymphocytes: PCS (High) | 0 | 1
  Neutrophils: PCS (Low) | 4 | 2
  Neutrophils: PCS (High) | 9 | 8
  Eosinophils: PCS (High) | 0 | 0
  Monocytes: PCS (High) | 0 | 0
  Basophils: PCS (High) | 0 | 0
  Direct Coombs test:- at Baseline, + post-Baseline | 15 | 2
  Hematocrit (ratio): PCS (Low) | 5 | 8
  Hematocrit (ratio): PCS (High) | 0 | 0

39. Secondary Outcome: Safety and Tolerability: Clinical Laboratory Evaluation Clinical Chemistry.
Description: Potentially clinically significant (PCS) post Baseline clinical chemistry values up to LFU (Safety analysis set)
Time Frame: study duration (from screening to Day 49 LFU visit)
Population: Safety analysis set: all patients who received at least 1 dose of IP
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 215 | 217
Number of patients
  Alanine aminotransferase (μkat/L): PCS (High) | 3 | 8
  Alkaline phosphatase (μkat/L): PCS (Low) | 0 | 0
  Alkaline phosphatase (μkat/L): PCS (High) | 2 | 3
  Aspartate aminotransferase (μkat/L): PCS (High) | 4 | 4
  Bicarbonate (mmol/L) PCS (Low) | 1 | 0
  Bicarbonate (mmol/L): PCS (High) | 0 | 0
  Creatinine (μmol/L): PCS (High) | 0 | 1
  Glucose (non-fasting) (mmol/L): PCS (Low) | 0 | 0
  Glucose (non-fasting) (mmol/L): PCS (High) | 1 | 1
  Gamma-glutamyl transferase (μkat/L):PCS (High) | 2 | 4
  Inorganic phosphorus (mmol/L): PCS (Low) | 3 | 7
  Inorganic phosphorus (mmol/L): PCS (High) | 0 | 0
  Potassium (mmol/L): PCS (Low) | 9 | 5
  Potassium (mmol/L): PCS (High) | 3 | 1
  Total bilirubin (μmol/L): PCS (High) | 0 | 1
  Direct bilirubin (μmol/L): PCS (High) | 1 | 1

40. Secondary Outcome: Safety and Tolerability:ECG , QTcB and QTcF Intervals
Description: Shifts in ECG interpretation and changes in QT, QTcB, and QTcF intervals , from baseline to post baseline.
Time Frame: EOT visit/any observation on treatment
Population: Safety analysis set: all patients who received at least 1 dose of IP
Measure: Number; unit: Number of patients
Arm/Group | Ceftazidime-Avibactam Plus Metronidazole | Meropenem
Number analyzed (Participants) | 215 | 217
Number of patients
  Normal to Abnormal: EOT | 17 | 14
  Normal to Abnormal: Anytime up to EOT | 34 | 30
  Reaching a value in QT: ≥450 (ms) | 9 | 10
  Reaching a value in QT: ≥480 (ms) | 2 | 1
  Reaching a value in QT: ≥500 (ms) | 0 | 0
  QT: ≥500 and increase from Baseline ≥60(ms) | 0 | 0
  Increase in QT: ≥30 (ms) | 115 | 114
  Increase in QT: ≥60 (ms) | 50 | 44
  Decrease in QT: ≥30 (ms) | 24 | 24
  Decrease in QT: ≥60 (ms) | 12 | 4
  Reaching a value in QTcB: ≥450(ms) | 57 | 63
  Reaching a value in QTcB: ≥480(ms) | 13 | 8
  Reaching a value in QTcB: ≥500 (ms) | 4 | 2
  QTcB: ≥500 and increase from Baseline ≥60(ms) | 2 | 1
  Increase in QTcB: ≥30 (ms) | 21 | 27
  Increase in QTcB: ≥60 (ms) | 2 | 1
  Decrease in QTcB: ≥30 (ms) | 42 | 26
  Decrease in QTcB: ≥60 (ms) | 6 | 4
  Reaching a value in QTcF: ≥450 (ms) | 19 | 18
  Reaching a value in QTcF: ≥480 (ms) | 4 | 0
  Reaching a value in QTcF: ≥500 (ms) | 1 | 0
  QTcF: ≥500 and increase from Baseline ≥60 (ms) | 0 | 0
  Increase in QTcF: ≥30 (ms) | 42 | 41
  Increase in QTcF: ≥60 (ms) | 4 | 3
  Decrease QTcF: ≥30 (ms) | 21 | 19
  Decrease QTcF: ≥60 (ms) | 7 | 1

41. Secondary Outcome: Plasma Concentrations for Ceftazidime and Avibactam
Description: Blood samples were taken from all patients on Day 3 for the pharmacokinetic evaluation of ceftazidime and avibactam plasma concentrations
Time Frame: At Day 3: Anytime within 15 minutes prior to or after stopping study drug, anytime between 30 and 90 minutes after stopping study drug, anytime between 300 minutes and 360 minutes after stopping study drug.
Population: PK analysis set
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Ceftazidime(1); Avibactam(1): 15 minutes before or after
- Ceftazidime(2); Avibactam(2): 30-90 minutes after
- Ceftazidime(3); Avibactam(3): 300-360 minutes after
Arm/Group | Ceftazidime(1) | Avibactam(1) | Ceftazidime(2) | Avibactam(2) | Ceftazidime(3) | Avibactam(3)
Number analyzed (Participants) | 195 | 195 | 193 | 193 | 192 | 192
ng/mL | 60300.4 [1390 to 1880000] | 10126.9 [197 to 435000] | 46473.9 [2080 to 210000] | 7289.3 [229 to 36300] | 9555.0 [1740 to 222000] | 1207.2 [227 to 36300]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the screening/consent visit until the late follow-up visit (i.e. Day -1/0 to Day 42). FOR SAE's - only those reported by 2 or more patients in either group are shown in this summary.
Description: AEs spontaneously reported by the patient or care provider or reported in response to the open question from the study center personnel, or revealed by observation were to be collected and recorded in the eCRF.
Arm/Group | CAZ-AVI Plus Metronidazole | Meropenem
Serious Adverse Events (participants affected / at risk) | 9/215 | 11/217
Other Adverse Events (participants affected / at risk) | 44/215 | 47/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI Plus Metronidazole (N=215) | Meropenem (N=217)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI Plus Metronidazole (N=215) | Meropenem (N=217)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 16 (20)
Nausea (Gastrointestinal disorders) | 18 (25) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (8) | 4 (5)
Pyrexia (General disorders) | 9 (12) | 12 (21)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to use such Confidential study information and not to disclose them to any other third parties, except that the undersigned shall not be prevented from using or disclosing information: (a) which by written records was previously known; (b) which is now public knowledge, (c) which is lawfully obtained by the undersigned from sources who have a lawful right to disclose such information.